CLINICAL TRIAL: NCT05081245
Title: A Randomized, Double-blind, Parallel Group, Placebo-controlled Study to Investigate the Efficacy, Safety, and Tolerability of ML-004 in Adolescents and Adults With Autism Spectrum Disorders (ASD).
Brief Title: ML-004 in Adolescents and Adults With Autism Spectrum Disorders (ASD)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MapLight Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ML-004-002
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD; Autism; Autism Spectrum Disorder; Social Communication
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Communication | interventions — Tablets

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized, double-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ML-004 (IR)/(ER) tablet (Experimental): ML-004 is a bilayer immediate-release (IR)/extended-release (ER, gastroretentive) oral tablet formulation. ML-004 is taken orally once daily and provided as a tablet in two dose strengths of 12 mg (3 mg IR/9 mg ER) and 24 mg tablet (6 mg IR/18 mg ER). Dose levels for this study are 12 mg (provided as one 12 mg tablet), 24 mg (one 24 mg tablet), 48 mg (two 24 mg tablets), and 72 mg (three 24 mg tablets).
  Interventions: Drug: ML-004 (IR)/(ER) tablet
- ML-004 Placebo (Placebo Comparator): Matched placebo oral tablets will consist of same excipients as the investigational drug but without any ML-004. Placebo taken orally once daily to match tablet number of ML-004 dose levels for 12 mg (1 tablet), 24 mg (1 tablet), 48 mg (2 tablets), and 72 mg (3 tablets).
  Interventions: Drug: ML-004 Placebo

INTERVENTIONS:
Drug: ML-004 (IR)/(ER) tablet — Participants will receive ML-004 once daily.
  Arms: ML-004 (IR)/(ER) tablet
Drug: ML-004 Placebo — Participants will receive matching placebo once daily.
  Arms: ML-004 Placebo

SUMMARY:
ML-004-002 is a multi-center, randomized, double-blind, parallel-group, placebo-controlled study that will enroll approximately 150 adolescent and adult subjects with ASD. The primary objective is to evaluate the efficacy of ML-004 compared with placebo in the improvement of social communication deficits in subjects with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 to 45 at screening
* Has a designated care/study partner who can reliably report on symptoms
* Has a diagnosis of Autism Spectrum Disorder (ASD)
* Has a body mass index (BMI) 18 through 34 kg/m², inclusive
* Full scale IQ (or equivalent) ≥55 score, with adequate verbal fluency, as determined by the Principal Investigator.
* Psychoactive medications and adjunctive therapies are stable for 4 weeks prior to screening
* Must be able to swallow study medication

Exclusion Criteria:

* Has Rett syndrome or Child Disintegrative Disorder
* Has participated in any other study and received any other investigational medication (other than COVID-19 vaccination) or device within 60 days prior to screening
* History of epilepsy without current adequate control, or any seizure in the 6 months preceding screening
* History of suicidal ideation or behavior in the past 12 months, or a positive response to C-SSRS questions 4 and/or 5
* Systolic blood pressure ≥140 mmHg (if adult) or >135 mmHg (if adolescent), or diastolic blood pressure ≥90 (if adult) or >85 mmHg (if adolescent), or a clinical history of uncontrolled or severe hypertension
* If female, is pregnant or lactating

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Autism Behavior Inventory (ABI)-Social Communication Domain Score | Baseline up to Day 110
  Change from baseline in the ABI-Social Communication Domain Score will be reported. The ABI is a 62-item questionnaire for reporting the behaviors of subjects (ages: 3 years-adulthood) diagnosed with ASD. The tool is suitable for completion by parents or care/study partners of people with ASD. Each item assesses either quality (from not at all to without help) or frequency (never to very often) of a particular behavior. The Social Communication domain score is the sum of the scores in the social communication domain divided by the number of items in the domain.

SECONDARY OUTCOMES:
Change from Baseline in Clinician Global Impression of Improvement (CGI-I) | Day 110
  The CGI-I score is a single-item instrument based on a 7-point scale routinely used in clinical trials to capture the Investigator's global impression of response. The Investigator or designee rates the improvement observed from 1 (very much improved) to 7 (very much worse).
Change from Baseline in Autism Behavior Inventory-Clinician (ABI-C) Score | Baseline up to Day 110
  The ABI-Clinician (ABI-C) captures the clinician rating of behaviors of a person with ASD that occurred over the week prior to assessment. It contains 14 items reflecting the core and associated autism behavior domains: Social Communication, Restrictive Behaviors, Mood and Anxiety, Self Regulation, and Challenging Behavior. Each item is rated on a 7-point scale from 1 (none; no symptoms present) to 7 (very severe; persistent interference with function or adaptation).
Change from Baseline in Aberrant Behavior Checklist 2-Irritability (ABC-I) Subscale Score | Baseline up to Day 110
  The ABC is a parent- or care/study partner-reported behavior rating assessment with five domains and 58 items, each rated on a 0 (not at all a problem) to 3 (the problem is severe in degree) scale. The irritability domain consists of 15 items.
Change from baseline in the Clinician Global Impression of Severity (CGI-S) Score | Baseline up to Day 110
  The CGI-S is a global assessment of the clinician-rater's impression of the severity of the participant's illness. It is rated on a scale of 1 (normal, not at all ill) to 7 (among the most extremely ill).
Change from baseline in the ABI Repetitive/Restrictive Behavior Domain Score | Baseline up to Day 110
  Each item on the ABI-Repetitive/Restrictive Behavior Domain is rated by frequency (never to very often). The domain score is the sum of all domain items scores divided by the number of items in the domain.
Change from baseline in the ABI Mood and Anxiety Domain Score | Baseline up to Day 110
  Each item on the ABI- Mood and Anxiety Domain is rated by frequency (never to very often). The domain score is the sum of all domain items scores divided by the number of items in the domain.
Change from baseline in the ABI Challenging Behavior Domain Score | Baseline up to Day 110
  Each item on the ABI- Challenging Behavior Domain is rated by frequency (never to very often). The domain score is the sum of all domain items scores divided by the number of items in the domain.
Change from baseline in the ABI Self-regulation Domain Score | Baseline up to Day 110
  Each item on the ABI- Self-regulation Domain is rated by frequency (never to very often). The domain score is the sum of all domain items scores divided by the number of items in the domain.
Change from baseline in the ABI-Short Form (ABI-S) Score | Baseline up to Day 110
  The ABI-S is a 24-item short version of the ABI, containing items from each of the five domains. The domain score for each domain is calculated as the sum of scores all domain items divided by the number of items in the domain.
Change from baseline in the ABC-Social Withdrawal (ABC-SW) Subscale Score | Baseline up to Day 110
  The ABC-SW subscale consists of 16 items of the ABC-2 rated from 0 (not at all a problem) to 3 (the problem is severe in degree).
Change from baseline in the Social Responsiveness Scale 2 (SRS-2) Score | Baseline up to Day 110
  The SRS-2 consists of 65 items across 5 subscales. Responses range from 1 (not true) to 4 (almost always true).
Change from baseline in the Vineland-3 (Domain Level Version) Score: total of Communication, Socialization, and Maladaptive behavior domains | Baseline up to Day 110
  The Vineland-3 Domain Level Version contains 5 domains. Responses on each item are rated from 0 (never) to 2 (usually).

CONTACTS AND LOCATIONS:
Locations (29):
- United States (24):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Southwest Autism Research & Resource Center, Clinical Research, Phoenix, Arizona
  - Cortica Healthcare, Glendale, California
  - NRC Research Institute, Orange, California
  - Cortica, San Rafael, California
  - Yale Child Study Center, New Haven, Connecticut
  - Children's National Health System - The Children's Research Institute (CRI), Washington D.C., District of Columbia
  - Abba Medical Group, Miami, Florida
  - APG Research, LLC, Orlando, Florida
  - University of South Florida Psychiatry and Behavioral Neurosciences, Tampa, Florida
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - University of Missouri, Thompson Center for Autism & Neurodevelopmental Disorders, Columbia, Missouri
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Nathan Kline Institute for Psychiatric Research, Orangeburg, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Center for Autism and the Developing Brain, New York State Psychiatric Institute, White Plains, New York
  - Ohio State University Nisonger Center, Columbus, Ohio
  - Suburban Research Associates, Media, Pennsylvania
  - BioBehavioral Research of Austin, Austin, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Road Runner Research, Ltd., San Antonio, Texas
  - Family Psychiatry of The Woodlands, The Woodlands, Texas
  - Cedar Clinical Research, Draper, Utah
  - Virginia Commonwealth University, Richmond, Virginia
- Australia (2):
  - Brain and Mind Centre, Camperdown, New South Wales
  - The Royal Children's Hospital, Murdoch Children's Research Institute, Parkville, Victoria
- Canada (3):
  - OCT Research ULC (dba Okanagan Clinical Trials), Kelowna, British Columbia
  - Lawson Health Research Institute/ London Health Sciences Centre, London, Ontario
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided